CLINICAL TRIAL: NCT05009758
Title: Moving Towards PREcision Medicine In United Airways Disease: Unraveling inflaMmatory Patterns in Asthmatic Patients With or Without Nasal Polyps (PREMIUM) - a Descriptive Pilot Study
Brief Title: Moving Towards Precision Medicine in United Airways Disease: Unraveling Inflammatory Patterns in Asthmatic Patients With or Without Nasal Polyps
Acronym: PREMIUM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Julia Eckl-Dorna, Ap. Prof. Priv.-Doz. Dr, Medical University of Vienna
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: PREMIUM2021
Record Dates: First submitted 2021-08-05; First posted 2021-08-17 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Asthma; Chronic Rhinosinusitis With Nasal Polyps; Chronic Rhinosinusitis (Diagnosis); Nasal Polyps
Keywords: Asthma; Chronic Rhinosinusitis (CRS); CRS with Nasal Polyps; CRS without Nasal Polyps; Inflammatory profile; Type 2 inflammation
MeSH Terms: conditions — Asthma; Disease; Nasal Polyps | interventions — Blood Specimen Collection; Bronchoscopy; Pregnancy Tests; Demography; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Subjects attending the outpatient clinic of the Department of Othorrinolaringology or Pulmonology of the Medical University of Vienna for symptoms of asthma or CRS with nasal polyposis will be recruited during their routine visit. After informing patients about the scopes of the study, they will be invited for a screening visit. During this visit, patients will be informed about the nature of the study and asked whether they are willing to participate. After signing the informed consent, they will undergo a screening visit to determine their eligibility for the study and group allotment. The following parameters will be recorded at the screening visit: medical history including concomitant medication, nasal examination (endoscopy), lung function and FeNO measurement, blood draw (eosinophil levels and for exploratory parameters). Thereafter, eligible patients will attend a single study visit for the collection of all clinical parameters and samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- T2-high asthma with nasal polyps (Active Comparator): * FeNO > 25 ppB
  * Had either two times >= 250 eosinophils /µl measured in the blood OR one measurement of blood eosinophils >= 250 cells/µl (one of the two measurements at the screening visit) and/or one measurement of sputum eosinophils > 2% within the last 12 months
  * Presence of CRSwNP as confirmed by endoscopy or CT according to the European Position Paper on Rhinosinusitis and CRSwNP Guidelines)
  * Patients with a history of treatment with monoclonal antibodies for asthma or polyps will only be included if at least a washout period of 5 half-lives or at least 3 months have passed
  Interventions: Procedure: Blood sampling; Procedure: Nasosorption; Procedure: Oral sampling; Procedure: Bronchoscopy; Procedure: Nasal biopsy; Procedure: Nasal sampling; Procedure: Nasal mucosa mRNA sampling; Diagnostic Test: Pregnancy test; Other: Medical history of patients, demographic data, concomitant medication, questionnaire; Diagnostic Test: UPSIT smell test; Procedure: Spirometry; Procedure: FeNO; Procedure: Lung X-Ray
- T2-high asthma without nasal polyps (Active Comparator): * FeNO > 25 ppB
  * Had either two times >= 250 eosinophils /µl measured in the blood OR one measurement of blood eosinophils >= 250 cells/µl (one of the two measurements at the screening visit) and/or one measurement of sputum eosinophils > 2% within the last 12 months
  * Absence of NP as confirmed by endoscopy or CT according to the European Position Paper on Rhinosinusitis and CRSwNP Guidelines)
  * Patients with a history of treatment with monoclonal antibodies for asthma or polyps will only be included if at least a washout period of 5 half-lives or at least 3 months have passed
  Interventions: Procedure: Blood sampling; Procedure: Nasosorption; Procedure: Oral sampling; Procedure: Bronchoscopy; Procedure: Nasal sampling; Procedure: Nasal mucosa mRNA sampling; Diagnostic Test: Pregnancy test; Other: Medical history of patients, demographic data, concomitant medication, questionnaire; Diagnostic Test: UPSIT smell test; Procedure: Spirometry; Procedure: FeNO; Procedure: Lung X-Ray
- CRSwNP in absence of asthma (Active Comparator): * Presence of CRSwNP as confirmed by endoscopy or CT according to the European Position Paper on Rhinosinusitis and Nasal Polyps Guidelines26
  * Evidence of Type 2 inflammation: blood eosinophils >= 250 cells/µl measured in the blood OR total IgE >100 kU/L26 at the screening visit
  * Absence of asthma and N-ERD
  * Patients with a history of treatment with monoclonal antibodies for asthma or polyps will only be included if at least a washout period of 5 half-lives or at least 3 months have passed
  Interventions: Procedure: Blood sampling; Procedure: Nasosorption; Procedure: Oral sampling; Procedure: Bronchoscopy; Procedure: Nasal biopsy; Procedure: Nasal sampling; Procedure: Nasal mucosa mRNA sampling; Diagnostic Test: Pregnancy test; Other: Medical history of patients, demographic data, concomitant medication, questionnaire; Diagnostic Test: UPSIT smell test; Procedure: Spirometry; Procedure: FeNO; Procedure: Lung X-Ray

INTERVENTIONS:
Procedure: Blood sampling — Blood collection for PBMC isolation, measurement of cytokines in serum, and mass cytometry
Procedure: Nasosorption — Nasosorptions will be applied for the collection of nasal secretions (Nasosorption FX-I, Hunt Developments (UK) Limited, Midhurst, West Sussex, United Kingdom). Under visualization, the device will be inserted into the nasal cavity and be placed along the lateral wall against the inferior turbinate. The index finger of the patient will be used to press onto the external aspects of the alar and lateral nasal cartilages to hold the device in place. After 1 minute, the devices will be removed.
Procedure: Oral sampling — For oral sampling, saliva collection devices (SuperSAL or PureSAL, Oasis Diagnostic Corporation, USA) will be applied followed by elution. Then swabs optimized for the collection of specimens will be applied (CLASSIQSwabs, Copan Diagnostics Inc. Murietta, CA, USA) to the dorsum of the tongue.
Procedure: Bronchoscopy — The bronchoscopy will be performed in the outpatient clinic of the Department of Pulmonology. Bronchial alveolar lavage (BAL): the bronchoscope is wedged in the segmental or subsegmental bronchus of the middle lobe. Up to 300 ml sterile normal saline is injected stepwise via handheld syringe and then gradually withdrawn back into the syringe. BAL fluid (BALF) will be prepared and further analyzed in the lab. Transbronchial biopsy (TBLB): performed by forceps in the lung periphery under fluoroscopy guidance. Up to 4 biopsies are taken in two different lobes of one lung with a distance of 1-2 cm to the pleura. TBLB is only performed in patients who have got not contraindications.
Procedure: Nasal biopsy — Nasal biopsies will be taken during routine endoscopy performed to score CRSwNP. Patients will receive local anesthesia and decongestants prior to obtaining the biopsy. Samples will either be embedded in OCT or processed for cellular analysis
  Arms: CRSwNP in absence of asthma; T2-high asthma with nasal polyps
Procedure: Nasal sampling — Swabs optimized for the collection of specimens will be applied (CLASSIQSwabs, Copan Diagnostics Inc. Murietta, CA, USA) to the anterior naris and middle meatus of each nostril
Procedure: Nasal mucosa mRNA sampling — Mucosal mRNA sampling will be performed using a 10cm nasal curette (either Rhino-Probe, Arlington Scientific, USA or Cellskim, Hunt Developments, UK). Under direct visualization, the curette will be brought to lie against the mid-inferior portion of the inferior turbinate. The curette will be pressed against the mucosal surface moved outwards 2-3 times. This motion will be repeated 2-3 times to ensure good sample collection. This curette and technique have been shown to cause no significant discomfort to patients and thus it has the advantage of no requirement for local anesthetics.
Diagnostic Test: Pregnancy test — In female patients, pregnancy will be excluded with a standard urine pregnancy test at the beginning of the main visit.
Other: Medical history of patients, demographic data, concomitant medication, questionnaire — Patients will be asked for their medical history including demographic data and concomitant medication. Details will be noted in the source data file. Furthermore, patients will receive a questionnaire including tools to assess QOL impairment by CRS and asthma
Diagnostic Test: UPSIT smell test — University of Pennsylvania Smell Identification Test (UPSIT) smell test will be performed by the patients during the study. It consists of 40 questions in 4 different booklets. The patient needs to scratch a sniff strip with the microencapsulated odorant using a pencil and mark his choice on four-choice multiple-choice questions. The test is then scored by the study team out of the 40 items.
Procedure: Spirometry — Lung function will be measured by spirometry in the lung function unit of the Department of Pulmonology. Spirometry will be performed according to American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines by authorized and properly certified personal.
Procedure: FeNO — Airway inflammation will be evaluated using a standardized single-breath FeNO test in accordance with the lung function unit of the Department of Pulmonology. A single exhalation technique recommended by the manufacturer will be followed. The FeNO measurements will not be performed within 2 weeks of a respiratory infection. The FeNO test will be performed prior to spirometry. Subjects should not eat or drink 1 hour prior to having the FeNO test. Subjects should not use their rescue SABA medication (e.g., albuterol/salbutamol) within 6 hours of the measurement. Inhaled bronchodilators (including ICS/LABA) should be withheld for the effect duration specific to the bronchodilator. If not, the assessment should be postponed till after the required time has passed since the meal or drink or bronchodilator inhalation. The NIOX VERO® Airway Inflammation Monitor will be used to measured FeNO in the lung function unit of the Department of Pulmonology.
Procedure: Lung X-Ray — After the bronchoscopy, a lung x-ray will be performed and patients will stay overnight in the ward of the Department of Pulmonology.

SUMMARY:
Asthma and chronic rhinosinusitis (CRS) are inflammatory diseases of the respiratory tract, asthma from the lower part, and CRS, from the upper part. In theory, these parts are correlated as if they are one single organ, namely "united airways", which means that if one is affected by any condition, the other might be impacted as well. However, this relationship has not yet been described down to the cellular and molecular levels. By investigating patients that have (1) asthma and CRS with nasal polyp, (2) asthma and CRS without nasal polyp, and (3) just CRS with nasal polyp, we aim to determine the correlation of the upper and lower part of the respiratory tract. At first, the characterization of disease will be determined by established clinical criteria, such as lung function, blood analysis for the presence of eosinophils (a type of white cells), and nasal polyp score. To continue, in-depth analysis of nose, oropharynx, and lung samples will help gain information about the inflammatory profile and local microbiome of the three different groups of patients through molecular and cellular assays. The results of this study will help to describe the hypothesis of the united airways which will provide better guidance for medical treatment of asthma and CRS with or without polyp, thus improving the life quality of patients.

DETAILED DESCRIPTION:
1. Background Both, asthma and chronic rhinosinusitis (CRS) are inflammatory conditions of the airways. The prevalence of asthma - with its cardinal symptoms wheezing, breathlessness, chest tightness, and coughing - has risen over the past decades not only in industrial but also in developing countries. For instance, about 8% of the United States' population and 8.2% of Europeans are diagnosed with asthma. Chronic rhinosinusitis with (CRSwNP) and without nasal polyps (CRSsNP) is a condition affecting up to 16% and 11% of the US and European population, respectively3. Both diseases, asthma and CRS, can severely impair quality of life as well as productivity and therefore embody an immense socioeconomic burden.

   Despite the distinction of the respiratory tract in the upper and lower airways, both parts are anatomically and immunologically related. This led to the concept of "United airway diseases" assuming that upper and lower airways form a single organ. Consequently, inflammation in the upper affects the lower respiratory tract and vice versa. This concept initially described in the context of allergic respiratory disease can also be extended to the link between sinonasal and lower airway diseases. Accordingly, the association between asthma and CRS prevalence has been unambiguously shown in epidemiological studies: around 20% of CRSsNP patients and around 48% of CRSwNP patients suffer from asthma. Conversely, nasal polyposis is detected in 19 to 25% of asthmatics. In cases of severe asthma, even up to 54% of patients were reported to have a history of nasal polyposis. However, the pathophysiological mechanism underlying the association of asthma and CRS has been poorly investigated so far.

   Based on the predominant inflammatory profile, asthma can be separated into T2-high and T2-low endotypes. Thereby, around 60% of severe asthma patients show a T2-high profile. The picture is becoming even more complex regarding classifications of CRS. Phenotypically we distinguish between CRSsNP and CRSwNP. However, up to 10 different endotypes of CRS can be defined based on various different inflammatory markers in nasal polyps or nasal secretions. Approaches to characterize endotypes describing conditions involving both asthma and CRS have barely been made so far.

   On a cellular and protein level, it seems that higher concentrations of Staphylococcus enterotoxin-specific IgE, total IgE and eosinophil cationic protein in nasal polyp tissue are indicators for a higher risk of asthma. Furthermore, it was observed that patients with CRS and eosinophilic asthma (as determined by FeNO levels only) show high numbers of eosinophils in their nasal polyps. This nasal polyp eosinophilia was associated with a more severe asthma phenotype as well as larger polyps and a significantly higher nasal polyp recurrence rate compared to non-eosinophilic patients. However, up to this point, no study investigated whether inflammatory profiles in polyps and asthmatic lungs correspond and how inflammatory profiles of patients suffering from asthma with or without polyps may differ.

   Novel antibody-based therapies targeting mediators of type 2 immune response are constantly emerging as new treatment options for patients with severe chronic airway diseases. Therapeutic antibodies targeting IgE or IL-4/IL-13, IL-5, or IL-5 receptor-mediated pathways are currently licensed for the treatment of asthma but have also successfully been used to treat CRSwNP to some extent. In this respect, anti-IgE (omalizumab) and anti-IL4α receptor (dupilumab) specific monoclonal antibodies have recently been licensed for the treatment of nasal polyps and CRSwNP respectively. Antibodies targeting molecules further upstream in the inflammatory cascade such as TSLP or IL-33 are currently under development. Anti-TSLP antibodies showed first promising results in clinical trials including patients suffering from uncontrolled asthma. Despite targeting molecular pathways involved in the pathogenesis of both diseases, some monoclonal antibodies such as reslizumab are effective in treating asthma but fail to significantly ameliorate nasal polyposis. Interestingly, a post-hoc responder analysis showed that the group of patients with high baseline IL-5 levels in nasal secretions improved upon reslizumab treatment, while the other patient groups did not. These findings illustrate the urgent need to better understand the pathomechanism and potential links underlying both diseases in order to choose the right therapy for the right patient.
2. Study rationale In this study, we aim to unravel the pathophysiological mechanisms underlying T2-high asthma with or without nasal polyposis. Therefore, we plan to thoroughly examine T2-high asthmatic patients with and without nasal polyposis at the cellular and molecular level and compare them to patients suffering from eosinophilic polyps in the absence of asthma. Deep analysis of nose, oropharynx, and lung samples will yield information on inflammatory patterns at protein and mRNA level, cellular tissue architecture in the different disease subtypes as well as microbiome composition. This pilot study will help to unravel underlying pathomechanisms in these united airway diseases and, therefore, provide a rationale for new therapy approaches including biologicals.
3. Study objectives

In this study we plan to:

* evaluate the inflammatory profile in different sections of the airways;
* evaluate the endotype and immunological profile of CRSwNP (when applicable);
* determine the microbiome composition in nose, oropharynx, and bronchi in T2-high asthmatic patients with and without CRSwNP, N-ERD compared to patients with CRSwNP in absence of asthma

ELIGIBILITY:
Inclusion Criteria:

All patients who

* 18-99 years of age
* have a recorded clinical diagnosis of asthma (ICD-10 Code: J45)
* undergo moderate-serve asthma treatment according to GINA/DAL treatment step 4 or step 5 without oral corticosteroid or monoclonal antibody therapy
* Asthma treatment for a minimum of 12 weeks prior to screening visit

  * Group 1 and 2 - T2-high asthma with or without polyps:
* FeNO > 25 ppB
* had either two times >= 250 eosinophils /µl measured in the blood OR one measurement of blood eosinophils >= 250 cells/µl (one of the two measurements at the screening visit) and/or one measurement of sputum eosinophils > 2% within the last 12 months
* Group with polyps: Presence of CRSwNP as confirmed by endoscopy or CT according to the European Position Paper on Rhinosinusitis and CRSwNP Guidelines)

  * Group 3 - CRSwNP in absence of asthma:
* Presence of CRSwNP as confirmed by endoscopy or CT according to the European Position Paper on Rhinosinusitis and Nasal Polyps Guidelines
* Evidence of Type 2 inflammation: eosinophils >= 250 cells/µl measured in the blood OR total IgE >100 kU/L at the screening visit
* Absence of asthma and N-ERD
* Patients with a history of treatment with monoclonal antibodies for asthma or polyps will only be included if at least a wash out period of 5 half-lives or at least 3 months have passed

Exclusion Criteria:

* Pregnancy (as determined by ß-HCG test)
* Patients with severe anatomic variations or deviations that do not allow access to all areas in the nasal cavity
* Patients undergoing chronic oral corticosteroid therapy
* Patients with any other confounding underlying lung disorder including but not limited to:

  * Bronchiectasis, chronic obstructive pulmonary disorder (COPD), pulmonary fibrosis, emphysema, primary ciliary dyskinesia
  * Cystic fibrosis, any known parasitic infections, and lung cancer
* Patients with pulmonary conditions with symptoms of asthma and blood eosinophilia including but not limited to: Eosinophilic granulomatosis with polyangiitis (EGPA), allergic bronchopulmonary aspergillus, and hypereosinophilic syndrome
* A mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Patients with clinically meaningful comorbidity as determined by the evaluating committee
* Patients with a history of exacerbation of chronic rhinosinusitis or asthma 4 weeks prior to any visit
* Intake of a burst of systemic corticosteroids 4 weeks prior to any visit.
* Immunosuppressive treatment (e.g. cyclosporine)
* Drug and alcohol abuses
* Current smoker
* Former smoker if stopped smoking <6 months and/or has >10 pack-years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Inflammatory profile in different sections of the airways | 2 years
  Concentration of selected inflammatory mediators in T2-high asthmatic patients with and without polyps and in patients with CRSwNP in absence of asthma

SECONDARY OUTCOMES:
Endotype and immunological profile of CRSwNP | 2 years
  Number of patients with specific endotypes of polyps and concentration of selected inflammatory mediators of various anatomic locations in the airways both in tissue and secretion samples in patients suffering from T2-high asthma with or without CRSwNP and in patients with CRSwNP in absence of asthma.
Microbiome composition in nose, oropharynx and bronchi in T2-high asthmatic patients with and without CRSwNP, N-ERD compared to patients with CRSwNP in absence of asthma | 2 years
  Number of different bacterial strains in different anatomical locations in asthmatic patients with and without polyps and CRSwNP patients in absence of asthma and to evaluate differences.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Eckl-Dorna, PhD, Principal Investigator — Medical University of Vienna; Sven Schneider, MD, Principal Investigator — Medical University of Vienna; Marco Idzko, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Allgemeines Krankenhaus (AKH) Wien, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stern J, Pier J, Litonjua AA. Asthma epidemiology and risk factors. Semin Immunopathol. 2020 Feb;42(1):5-15. doi: 10.1007/s00281-020-00785-1. Epub 2020 Feb 4. PMID 32020334
- [Background] Gibson GJ, Loddenkemper R, Lundback B, Sibille Y. Respiratory health and disease in Europe: the new European Lung White Book. Eur Respir J. 2013 Sep;42(3):559-63. doi: 10.1183/09031936.00105513. No abstract available. PMID 24000245
- [Background] Hellings PW, Klimek L, Cingi C, Agache I, Akdis C, Bachert C, Bousquet J, Demoly P, Gevaert P, Hox V, Hupin C, Kalogjera L, Manole F, Mosges R, Mullol J, Muluk NB, Muraro A, Papadopoulos N, Pawankar R, Rondon C, Rundenko M, Seys SF, Toskala E, Van Gerven L, Zhang L, Zhang N, Fokkens WJ. Non-allergic rhinitis: Position paper of the European Academy of Allergy and Clinical Immunology. Allergy. 2017 Nov;72(11):1657-1665. doi: 10.1111/all.13200. Epub 2017 Jun 2. PMID 28474799
- [Background] Loftus PA, Wise SK. Epidemiology and economic burden of asthma. Int Forum Allergy Rhinol. 2015 Sep;5 Suppl 1:S7-10. doi: 10.1002/alr.21547. Epub 2015 May 23. PMID 26010063
- [Background] Smith KA, Orlandi RR, Rudmik L. Cost of adult chronic rhinosinusitis: A systematic review. Laryngoscope. 2015 Jul;125(7):1547-56. doi: 10.1002/lary.25180. Epub 2015 Jan 30. PMID 25640115
- [Background] Giavina-Bianchi P, Aun MV, Takejima P, Kalil J, Agondi RC. United airway disease: current perspectives. J Asthma Allergy. 2016 May 11;9:93-100. doi: 10.2147/JAA.S81541. eCollection 2016. PMID 27257389
- [Background] Passalacqua G, Ciprandi G, Canonica GW. United airways disease: therapeutic aspects. Thorax. 2000 Oct;55 Suppl 2(Suppl 2):S26-7. doi: 10.1136/thorax.55.suppl_2.s26. No abstract available. PMID 10992552
- [Background] Yii ACA, Tay TR, Choo XN, Koh MSY, Tee AKH, Wang DY. Precision medicine in united airways disease: A "treatable traits" approach. Allergy. 2018 Oct;73(10):1964-1978. doi: 10.1111/all.13496. Epub 2018 Jul 10. PMID 29869791
- [Background] Promsopa C, Kansara S, Citardi MJ, Fakhri S, Porter P, Luong A. Prevalence of confirmed asthma varies in chronic rhinosinusitis subtypes. Int Forum Allergy Rhinol. 2016 Apr;6(4):373-7. doi: 10.1002/alr.21674. Epub 2015 Dec 17. PMID 26678021
- [Background] Philpott CM, Erskine S, Hopkins C, Kumar N, Anari S, Kara N, Sunkaraneni S, Ray J, Clark A, Wilson A; CRES group; Erskine S, Philpott C, Clark A, Hopkins C, Robertson A, Ahmed S, Kara N, Carrie S, Sunkaraneni V, Ray J, Anari S, Jervis P, Panesaar J, Farboud A, Kumar N, Cathcart R, Almeyda R, Khalil H, Prinsley P, Mansell N, Salam M, Hobson J, Woods J, Coombes E. Prevalence of asthma, aspirin sensitivity and allergy in chronic rhinosinusitis: data from the UK National Chronic Rhinosinusitis Epidemiology Study. Respir Res. 2018 Jun 27;19(1):129. doi: 10.1186/s12931-018-0823-y. PMID 29945606
- [Background] Ahmadiafshar A, Farjd HR, Moezzi F, Mousavinasab N. Nasal polyposis in patients with asthma and allergic rhinitis. J Laryngol Otol. 2012 Aug;126(8):780-3. doi: 10.1017/S0022215112000771. Epub 2012 Jun 12. PMID 22691577
- [Background] de Groot JC, Storm H, Amelink M, de Nijs SB, Eichhorn E, Reitsma BH, Bel EH, Ten Brinke A. Clinical profile of patients with adult-onset eosinophilic asthma. ERJ Open Res. 2016 May 26;2(2):00100-2015. doi: 10.1183/23120541.00100-2015. eCollection 2016 Apr. PMID 27730197
- [Background] Amelink M, de Groot JC, de Nijs SB, Lutter R, Zwinderman AH, Sterk PJ, ten Brinke A, Bel EH. Severe adult-onset asthma: A distinct phenotype. J Allergy Clin Immunol. 2013 Aug;132(2):336-41. doi: 10.1016/j.jaci.2013.04.052. Epub 2013 Jun 24. PMID 23806634
- [Background] Narendra D, Blixt J, Hanania NA. Immunological biomarkers in severe asthma. Semin Immunol. 2019 Dec;46:101332. doi: 10.1016/j.smim.2019.101332. Epub 2019 Nov 14. PMID 31735516
- [Background] Tomassen P, Vandeplas G, Van Zele T, Cardell LO, Arebro J, Olze H, Forster-Ruhrmann U, Kowalski ML, Olszewska-Ziaber A, Holtappels G, De Ruyck N, Wang X, Van Drunen C, Mullol J, Hellings P, Hox V, Toskala E, Scadding G, Lund V, Zhang L, Fokkens W, Bachert C. Inflammatory endotypes of chronic rhinosinusitis based on cluster analysis of biomarkers. J Allergy Clin Immunol. 2016 May;137(5):1449-1456.e4. doi: 10.1016/j.jaci.2015.12.1324. Epub 2016 Mar 4. PMID 26949058
- [Background] Turner JH, Chandra RK, Li P, Bonnet K, Schlundt DG. Identification of clinically relevant chronic rhinosinusitis endotypes using cluster analysis of mucus cytokines. J Allergy Clin Immunol. 2018 May;141(5):1895-1897.e7. doi: 10.1016/j.jaci.2018.02.002. Epub 2018 Feb 13. No abstract available. PMID 29452200
- [Background] Bachert C, Zhang N, Holtappels G, De Lobel L, van Cauwenberge P, Liu S, Lin P, Bousquet J, Van Steen K. Presence of IL-5 protein and IgE antibodies to staphylococcal enterotoxins in nasal polyps is associated with comorbid asthma. J Allergy Clin Immunol. 2010 Nov;126(5):962-8, 968.e1-6. doi: 10.1016/j.jaci.2010.07.007. PMID 20810157
- [Background] Wu D, Li L, Zhang M, Wang J, Wei Y. Two inflammatory phenotypes of nasal polyps and comorbid asthma. Ann Allergy Asthma Immunol. 2017 Mar;118(3):318-325. doi: 10.1016/j.anai.2016.12.018. Epub 2017 Jan 23. PMID 28126433
- [Background] Fokkens WJ, Lund V, Bachert C, Mullol J, Bjermer L, Bousquet J, Canonica GW, Deneyer L, Desrosiers M, Diamant Z, Han J, Heffler E, Hopkins C, Jankowski R, Joos G, Knill A, Lee J, Lee SE, Marien G, Pugin B, Senior B, Seys SF, Hellings PW. EUFOREA consensus on biologics for CRSwNP with or without asthma. Allergy. 2019 Dec;74(12):2312-2319. doi: 10.1111/all.13875. Epub 2019 Jul 15. PMID 31090937
- [Background] Agache I, Rocha C, Beltran J, Song Y, Posso M, Sola I, Alonso-Coello P, Akdis C, Akdis M, Canonica GW, Casale T, Chivato T, Corren J, Del Giacco S, Eiwegger T, Firinu D, Gern JE, Hamelmann E, Hanania N, Makela M, Martin IH, Nair P, O'Mahony L, Papadopoulos NG, Papi A, Park HS, Perez de Llano L, Quirce S, Sastre J, Shamji M, Schwarze J, Canelo-Aybar C, Palomares O, Jutel M. Efficacy and safety of treatment with biologicals (benralizumab, dupilumab and omalizumab) for severe allergic asthma: A systematic review for the EAACI Guidelines - recommendations on the use of biologicals in severe asthma. Allergy. 2020 May;75(5):1043-1057. doi: 10.1111/all.14235. PMID 32064642
- [Background] Agarwal A, Spath D, Sherris DA, Kita H, Ponikau JU. Therapeutic Antibodies for Nasal Polyposis Treatment: Where Are We Headed? Clin Rev Allergy Immunol. 2020 Oct;59(2):141-149. doi: 10.1007/s12016-019-08734-z. PMID 31073812
- [Background] Han JK, Bachert C, Fokkens W, Desrosiers M, Wagenmann M, Lee SE, Smith SG, Martin N, Mayer B, Yancey SW, Sousa AR, Chan R, Hopkins C; SYNAPSE study investigators. Mepolizumab for chronic rhinosinusitis with nasal polyps (SYNAPSE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Respir Med. 2021 Oct;9(10):1141-1153. doi: 10.1016/S2213-2600(21)00097-7. Epub 2021 Apr 16. PMID 33872587
- [Background] Agache I, Cojanu C, Laculiceanu A, Rogozea L. Critical Points on the Use of Biologicals in Allergic Diseases and Asthma. Allergy Asthma Immunol Res. 2020 Jan;12(1):24-41. doi: 10.4168/aair.2020.12.1.24. PMID 31743962
- [Background] Corren J, Parnes JR, Wang L, Mo M, Roseti SL, Griffiths JM, van der Merwe R. Tezepelumab in Adults with Uncontrolled Asthma. N Engl J Med. 2017 Sep 7;377(10):936-946. doi: 10.1056/NEJMoa1704064. PMID 28877011
- [Background] Gevaert P, Lang-Loidolt D, Lackner A, Stammberger H, Staudinger H, Van Zele T, Holtappels G, Tavernier J, van Cauwenberge P, Bachert C. Nasal IL-5 levels determine the response to anti-IL-5 treatment in patients with nasal polyps. J Allergy Clin Immunol. 2006 Nov;118(5):1133-41. doi: 10.1016/j.jaci.2006.05.031. Epub 2006 Sep 26. PMID 17088140
- [Background] Fokkens W, Lund V, Bachert C, Clement P, Helllings P, Holmstrom M, Jones N, Kalogjera L, Kennedy D, Kowalski M, Malmberg H, Mullol J, Passali D, Stammberger H, Stierna P; EAACI. EAACI position paper on rhinosinusitis and nasal polyps executive summary. Allergy. 2005 May;60(5):583-601. doi: 10.1111/j.1398-9995.2005.00830.x. No abstract available. PMID 15813802
- [Background] Meltzer EO, Hamilos DL, Hadley JA, Lanza DC, Marple BF, Nicklas RA, Adinoff AD, Bachert C, Borish L, Chinchilli VM, Danzig MR, Ferguson BJ, Fokkens WJ, Jenkins SG, Lund VJ, Mafee MF, Naclerio RM, Pawankar R, Ponikau JU, Schubert MS, Slavin RG, Stewart MG, Togias A, Wald ER, Winther B; Rhinosinusitis Initiative. Rhinosinusitis: developing guidance for clinical trials. J Allergy Clin Immunol. 2006 Nov;118(5 Suppl):S17-61. doi: 10.1016/j.jaci.2006.09.005. PMID 17084217
- [Background] Leaker BR, Malkov VA, Mogg R, Ruddy MK, Nicholson GC, Tan AJ, Tribouley C, Chen G, De Lepeleire I, Calder NA, Chung H, Lavender P, Carayannopoulos LN, Hansel TT. The nasal mucosal late allergic reaction to grass pollen involves type 2 inflammation (IL-5 and IL-13), the inflammasome (IL-1beta), and complement. Mucosal Immunol. 2017 Mar;10(2):408-420. doi: 10.1038/mi.2016.74. Epub 2016 Sep 28. PMID 27677865
- [Background] Yan M, Pamp SJ, Fukuyama J, Hwang PH, Cho DY, Holmes S, Relman DA. Nasal microenvironments and interspecific interactions influence nasal microbiota complexity and S. aureus carriage. Cell Host Microbe. 2013 Dec 11;14(6):631-40. doi: 10.1016/j.chom.2013.11.005. PMID 24331461
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675
- [Background] Callahan BJ, McMurdie PJ, Rosen MJ, Han AW, Johnson AJ, Holmes SP. DADA2: High-resolution sample inference from Illumina amplicon data. Nat Methods. 2016 Jul;13(7):581-3. doi: 10.1038/nmeth.3869. Epub 2016 May 23. PMID 27214047
- [Background] Pruesse E, Peplies J, Glockner FO. SINA: accurate high-throughput multiple sequence alignment of ribosomal RNA genes. Bioinformatics. 2012 Jul 15;28(14):1823-9. doi: 10.1093/bioinformatics/bts252. Epub 2012 May 3. PMID 22556368
- [Background] Quast C, Pruesse E, Yilmaz P, Gerken J, Schweer T, Yarza P, Peplies J, Glockner FO. The SILVA ribosomal RNA gene database project: improved data processing and web-based tools. Nucleic Acids Res. 2013 Jan;41(Database issue):D590-6. doi: 10.1093/nar/gks1219. Epub 2012 Nov 28. PMID 23193283
- [Background] Davis NM, Proctor DM, Holmes SP, Relman DA, Callahan BJ. Simple statistical identification and removal of contaminant sequences in marker-gene and metagenomics data. Microbiome. 2018 Dec 17;6(1):226. doi: 10.1186/s40168-018-0605-2. PMID 30558668
- [Background] Wilson N, Zhao N, Zhan X, Koh H, Fu W, Chen J, Li H, Wu MC, Plantinga AM. MiRKAT: kernel machine regression-based global association tests for the microbiome. Bioinformatics. 2021 Jul 12;37(11):1595-1597. doi: 10.1093/bioinformatics/btaa951. PMID 33225342
- [Background] Love MI, Huber W, Anders S. Moderated estimation of fold change and dispersion for RNA-seq data with DESeq2. Genome Biol. 2014;15(12):550. doi: 10.1186/s13059-014-0550-8. PMID 25516281
- [Background] Le Cao KA, Costello ME, Lakis VA, Bartolo F, Chua XY, Brazeilles R, Rondeau P. MixMC: A Multivariate Statistical Framework to Gain Insight into Microbial Communities. PLoS One. 2016 Aug 11;11(8):e0160169. doi: 10.1371/journal.pone.0160169. eCollection 2016. PMID 27513472
- [Background] Alving, K., Anolik, R., Crater, G. et al. Validation of a New Portable Exhaled Nitric Oxide Analyzer, NIOX VERO®: Randomized Studies in Asthma. Pulm Ther 3, 207-218 (2017). https://doi.org/10.1007/s41030-017-0032-8